CLINICAL TRIAL: NCT04650074
Title: Pilot Study to Evaluate the Effectiveness of a Mixture of Ketamine / Lidocaine Administered by Mesotherapy in the Management of Neuropathic Pain in Complex Regional Pain Syndrome Type 1 (CRPS1). A Monocentric Randomized and Controlled Clinical Study
Brief Title: Effectiveness of Ketamine Administered by Mesotherapy in Complex Regional Pain Syndrome Type 1 (CRPS1)
Acronym: MESO-SDRC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 69HCL18_0996
Record Dates: First submitted 2020-11-25; First posted 2020-12-02 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Neuropathic Pain; Complex Regional Pain Syndrome Type 1
Keywords: Complex Regional Pain Syndrome Type 1; Mesotherapy; Lidocaïne; Ketamine; Randomized clinical trial
MeSH Terms: conditions — Neuralgia; Complex Regional Pain Syndromes | interventions — Lidocaine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LIDOCAINE 20 mg (Active Comparator): 4 injections (on day 1, day 7, day 14, day 28) by mesotherapy of 20 mg Lidocaine (qsp 6 ml NaCl 0.9%).
  Interventions: Drug: LIDOCAINE 20 mg
- LIDOCAINE 20 mg + KETAMINE 20 mg (Experimental): 4 injections (on day 1, day 7, day 14, day 28) by mesotherapy of 20 mg Lidocaine + 20 mg Ketamine (qsp 6 ml NaCl 0.9%).
  Interventions: Drug: LIDOCAINE 20 mg + KETAMINE 20 mg
- LIDOCAINE 20 mg + KETAMINE 40 mg (Experimental): 4 injections (on day 1, day 7, day 14, day 28) by mesotherapy of 20 mg Lidocaine + 40 mg Ketamine (qsp 6 ml NaCl 0.9%).
  Interventions: Drug: LIDOCAINE 20 mg + KETAMINE 40 mg

INTERVENTIONS:
Drug: LIDOCAINE 20 mg — 4 injections (on day 1, day 7, day 14, day 28) by mesotherapy of 20 mg Lidocaine (qsp 6 ml NaCl 0.9%).
  Each mesotherapy session includes 2 steps performed chronologically. It will be done within 2 or 3 minutes each one:
  * 1st sequence: intra-epidermal injections of 3 ml by manual technique in crossed lines with a 13 mm x 0.30 needle,
  * 2nd sequence : superficial intradermal injections of 3 ml (between 1 and 2 mm) using a technique assisted by a Pistor Eliance injector at a frequency of 200 punctures per minute.
  Arms: LIDOCAINE 20 mg
Drug: LIDOCAINE 20 mg + KETAMINE 20 mg — 4 injections (on day 1, day 7, day 14, day 28) by mesotherapy of 20 mg Lidocaine + 20 mg Ketamine (qsp 6 ml NaCl 0.9%).
  Each mesotherapy session includes 2 steps performed chronologically. It will be done within 2 or 3 minutes each one:
  * 1st sequence: intra-epidermal injections of 3 ml by manual technique in crossed lines with a 13 mm x 0.30 needle,
  * 2nd sequence : superficial intradermal injections of 3 ml (between 1 and 2 mm) using a technique assisted by a Pistor Eliance injector at a frequency of 200 punctures per minute.
  Arms: LIDOCAINE 20 mg + KETAMINE 20 mg
Drug: LIDOCAINE 20 mg + KETAMINE 40 mg — 4 injections (on day 1, day 7, day 14, day 28) by mesotherapy of 20 mg Lidocaine + 40 mg Ketamine (qsp 6 ml NaCl 0.9%).
  Each mesotherapy session includes 2 steps performed chronologically. It will be done within 2 or 3 minutes each one:
  * 1st sequence: intra-epidermal injections of 3 ml by manual technique in crossed lines with a 13 mm x 0.30 needle,
  * 2nd sequence : superficial intradermal injections of 3 ml (between 1 and 2 mm) using a technique assisted by a Pistor Eliance injector at a frequency of 200 punctures per minute
  Arms: LIDOCAINE 20 mg + KETAMINE 40 mg

SUMMARY:
Complex Regional Pain Syndrome type 1 (CRPS1) is a disabling pain syndrome. Its definitive treatment has not been established and the results of current treatments are often unsatisfactory.

The prognosis is difficult to establish because the vast majority of CRPS regresses within a few weeks. However, some forms are hyperalgesic with a major chronic painful picture, very debilitating and responding poorly to treatments with possible permanent sequelae.

The management of CRPS remains difficult and unsatisfactory and is symptomatic, multidimensional and multidisciplinary involving medical, paramedical and socio-professional workers. The priority therapeutic objectives are analgesia, maintenance or gain of joint range and maintenance or restoration of motor functions. This treatment is not the subject of a consensus and its implementation is sometimes the responsibility of specialized centers such as "pain relief" centers or even Physical Medicine and Rehabilitation (MPR) structures.

Previous studies using ketamine as a treatment for CRPS1 show encouraging results with a decrease in neuropathic pain. Ketamine is a low dose pain reliever. Ketamine has been studied as an adjuvant for the treatment of chronic pain, particularly neuropathic pain. The results suggest that ketamine decreases pain intensity and reduces opioid reliance when used as an adjunct to chronic and acute pain. Ketamine is believed to have a greater analgesic effect in patients with CRPS1 compared to other chronic pain syndromes. In these studies, ketamine was used intravenously, subcutaneously, orally, intranasally, or topically.

Mesotherapy allows microdose local treatment to be carried out limiting side effects, ensuring compliance and easy to implement. The injected solutions often contain a local anesthetic (procaine or lidocaine). It allows better local tolerance from the start of treatment. In addition, through its vasodilator effect on the microcirculation, it increases the effectiveness and tolerance of other injected products.

There are no studies using ketamine administrated by mesotherapy. Based on the scientific literature, there are good reasons to believe that this treatment could be effective on the neuropathic pain of CRPS1 and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Male / female aged ≥18 years,
* Patient suffering from Complex Regional Pain Syndrome Type 1 (CRPS1), according to the Budapest criteria, with a neuropathic component limited to the lower or upper limbs diagnosed by the Neuropathic pain DN4 Questionnaire
* Patient having undergone a three-stage dynamic bone scan less than 3 months old : vascular, tissue, bone, showing diffuse and extensive hyperfixation in the area suspected of CRPS1,
* Negative urinary pregnancy test in women of childbearing age,
* VAS (Visual Analogue Scale) > 50mm (on a scale of 0 to 100 mm) at inclusion,
* Patients affiliated to the French social security system,
* Writing informed consent obtained.

Exclusion Criteria:

* Patient with the following medical history or ongoing pathologies: epilepsy, hypertension (> 180mm / 100mm Hg), unbalanced coronary artery disease, recent myocardial infarction (MDI) (less than 12 months), porphyria, hyperthyroidism, known Behçet's disease, known blood crass disorder or PT (Prothrombin Time) <20%, known psychiatric disorders, known septic osteoarticular disease,
* Patient with HIV ((Human Immunodeficiency Viruses) infection, immunosuppression and / or immunosuppressive treatment
* Severe heart failure,
* History of severe allergy (angioedema),
* Known allergies to Cr and Zn,
* Current skin infection,
* Skin lesion next to the injection area
* Phobia of injections,
* Known hypersensitivity to ketamine hydrochloride or chlorobutanol,
* Known hypersensitivity to lidocaine hydrochloride or to amide-linked local anesthetics,
* Pregnant or breastfeeding woman
* Patient under protective measure (safeguard measure, curatorship, guardianship) or deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) score | On day 0 (inclusion) and day 56 (end of patient follow-up)
  Pain measured by VAS (Visual Analogue Scale)

SECONDARY OUTCOMES:
Evolution of the Visual Analogue Scale score | On day 0 (inclusion), on day 1, day 7, day 14 and day 28 (mesotherapy sessions), and on day 56 (end of patient follow-up)
  The VAS (Visual Analogue Scale) score will be assessed at inclusion, before each mesotherapy session, and at the end of the patient follow-up
Neuropathic Pain Symptom Inventory (NPSI) self-questionnaire score | On day 0 (inclusion), on day 1, day 7, day 14 and day 28 (mesotherapy sessions), and on day 56 (end of the patient follow-up)
  The Neuropathic pain will be assessed using the NPSI (Neuropathic Pain Symptom Inventory self-questionnaire) at inclusion, before each mesotherapy session, and at the patients withdrawal.
Brief Pain Inventory (BPI) self-questionnaire score | On day 0 (inclusion) and on day 56 (end of patient follouw-up)
  The main dimensions of pain (i.e. intensity, functional disability, social and family repercussions as well as the level of psychological distress) will be assessed using the BPI (Brief Pain Inventory self-questionnaire) at inclusion and at the patients withdrawal.
Relevant adverse events | Until day 56 (end of patient follow-up)
  The relevant adverse events (AEs), as well as the average of the highest grades of the relevant adverse events, will be collected during the patient follow-up, in particular after each mesotherapy session. The physician will ask the patient at each of the visits and will report any adverse event (AE). The nature and intensity of the AE will be assessed according to the Common Terminology Criteria for Adverse Events grid (CTCAE version 5.0). Relevant adverse events (AEs at least possibly related to treatment or mesotherapy) will be considered.
Concomitant consumption of analgesics | Until day 56 (end of patient follow-up)
  The consumption of other analgesics concomitant with the treatment will be recorded
EQ-5D-5L (EuroQol health states) questionnaire score | On day 1 (inclusion) and on day 56 (end of patient follow-up)
  The quality of life will be assessed using the EQ-5D-5L questionnaire (EuroQol health states)
Visual Analogue Scale and Adverse Events grades (Benefit / risk balance) | Until day 56 (end of patient follow-up)
  To simultaneously compare the VAS (Visual Analogue Scale) and the relevant adverse events (AE) grades between groups.
  This benefit-risk balance will be estimate in a hierarchical fashion using the method of pairwise comparisons. The VAS will be used as the first endpoint (benefit) and the highest grade of AE in a given patient as the second endpoint (risk). No clinical relevance threshold will be specified for the two criteria for the primary analysis, but they will then be added as a sensitivity analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of orthopedic surgery and trauma emergencies of the lower limb, Edouard Herriot Hospital, Hospices Civils de Lyon, Lyon, France